CLINICAL TRIAL: NCT05213429
Title: Middle East Coronary Artery Ectasia Registry (MECAER): Incidence, Management, and One-Year Prognosis: A Multi-Centre Prospective Cohort Study.
Brief Title: Middle East Coronary Artery Ectasia Registry
Acronym: MECAER
Status: Recruiting | Type: Observational
Sponsor: Jordanian Research and Artificial Intelligence Group (Other)
Responsible Party: Sponsor
Other Study IDs: JoRAI group
Record Dates: First submitted 2022-01-04; First posted 2022-01-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: non interventional study — non interventional

SUMMARY:
This research project is the first in Jordan and Middle East in providing detailed registration of coronary ectasia cases provided by their primary healthcare providers. The investigators responsible for conducting this research are physicians and their teams who deal with patients with coronary ectasia in their clinics including the public and private medical sectors.

DETAILED DESCRIPTION:
Coronary artery ectasia (CAE) is the diffuse dilatation of coronary artery. It is defined as a dilatation with a diameter of 1.5 times the adjacent normal coronary artery. Its prevalence ranges from 1.2%-4.9% with male to female ratio of 3:1 .

Coronary ectasia likely represents an exaggerated form of expansive vascular remodeling (i.e. excessive expansive remodeling) in response to atherosclerotic plaque growth .

CAE is more common in males. Hypertension is a risk Factor. Interestingly, patients with DM have low incidence of CAE. This may be due to down regulation of MMP with negative remodeling in response to atherosclerosis . Smoking appears to be more common in patients with CAE than in those with coronary artery disease (CAD).

The angiographic classification for CAE (described by Markis et al.) categorizes the severity based on the extent of coronary arterial involvement: Type 1: Diffuse ectasia of 2-3 arteries; Type 2: Diffuse ectasia in one artery and localized in another; Type 3: Diffuse single arterial ectasia; Type 4: Localized or segmental ectasia.

Stable angina is the most common presentation in patients with CAE . Patients with CAE without stenosis had positive results during treadmill exercise tests. ST-elevation myocardial infarction (MI) , non-ST elevation MI can occur from altered blood flow by distal embolization or occlusion of ectatic segment with thrombus.

Medical management for CAE is a controversial area as there is lack of evidence based medicine, especially the role of antiplatelet versus anticoagulant agents. Aspirin was suggested in all patients because of coexistence of CAE with obstructive coronary lesions in the great majority of patients and the observed incidence of myocardial infarction, even in patients with isolated coronary ectasia .The role of dual anti platelet therapy has not been evaluated in prospective randomized studies. Based on the significant flow disturbances within the ecstatic segments, chronic anticoagulation with warfarin as main therapy was suggested

this study aims to fill the existing gap in the cardiac community about the topic of coronary ectasia. There is a substantial lack of dependable scientific data regarding the prevalence and disease prognosis of coronary ectasia. Screening, management and follow-up of coronary ectasia patients combined with comparative tests with reference studies will be initiated. A direct impact on improving coronary ectasia prognostic outcomes is expected by focusing efforts on determining the prevalence, prognosis and management procedures of ectasia. collected data will aid in improving the current therapeutic approaches to coronary ectasia and providing better control and management of coronary ectasia cases in the Middle East.

Study objectives:

Taking into account the classical coronary ectasia definition, the investigators propose:

* ANATOMIC OBJECTIVES.

  * To characterize coronary ectasia prevalence causing invasive coronary angiography.
  * To describe anatomy, location and aneurysms features.
  * To assess intracoronary imaging data if available.
  * To determine the underlying causes of coronary ectasia in patients
* CLINICAL OBJECTIVES.

  * Determine the cause for the diagnostic catheterization and ectasia symptoms, if present.
  * Patient´s clinical features.
  * Long-term outcomes.
* THERAPEUTIC OBJECTIVES.

  * To assess management strategies (conservative, interventional or surgical) and its short and long term results.
  * Disease management outcomes .

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected CAD who are referred for elective coronary angiography and fit the Coronary ectasia definition.

Exclusion Criteria:

* Patient younger than 18 years old.
* Patients who refuse to sign a consent form . Patients who are enrolled in another Ectasia study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a coronary Ectasia diagnosis after PCI imaging
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 1 year
  MI, stroke, angina and hospitalization

SECONDARY OUTCOMES:
all cause of death | 1 year
  CV death , Non-CV death

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud I Izraiq, MD, FACC, FSCAI, Study Chair — Jordanian Research and Artificial Intelligence Group
Locations (1):
- Specialty Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devabhaktuni S, Mercedes A, Diep J, Ahsan C. Coronary Artery Ectasia-A Review of Current Literature. Curr Cardiol Rev. 2016;12(4):318-323. doi: 10.2174/1573403x12666160504100159. PMID 27142049
- [Background] Hartnell GG, Parnell BM, Pridie RB. Coronary artery ectasia. Its prevalence and clinical significance in 4993 patients. Br Heart J. 1985 Oct;54(4):392-5. doi: 10.1136/hrt.54.4.392. PMID 4052280
- [Background] Willner NA, Ehrenberg S, Musallam A, Roguin A. Coronary artery ectasia: prevalence, angiographic characteristics and clinical outcome. Open Heart. 2020 Apr;7(1):e001096. doi: 10.1136/openhrt-2019-001096. PMID 32515749